CLINICAL TRIAL: NCT06915610
Title: Reengineering Cervical Cancer Screening for the 21st Century: Joint Action for a Novel Up-to-date and Sustainable Screening Program
Acronym: JANUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Saude Publica da Universidade do Porto (Other)
Collaborators: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other); Universidade do Porto (Other); Unidade Local de Saude de Gaia e Espinho EPE (Other)
Responsible Party: Principal Investigator, Nuno Lunet, Professor, Instituto de Saude Publica da Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MPr-2023-12-15422
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer Screening
Keywords: Cervical cancer; Human papillomavirus; Self-sampling; DNA methylation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Within each group, participants will be initially invited for CCS though one of the methods under evaluation, and those not adhering will be invited again for CCS through another method. This design will allow for between-group comparisons, both after the first invitation and considering the two invitations, as well as within-group comparisons to assess the extent to which the second (complementary) invitation may contribute to improve participation in CCS. Additionally, data on the participation in CCS in the same settings in the previous years will be retrospectively collected, allowing further ("before-after") comparisons within each group.
  A qualitative study will be conducted involving medical doctors and females invited for CCS within the study to assess barriers and facilitators to CCS implementation and participation.
  An observational design nested within the RCT will be used to assess the experience of females invited for CCS, and determinants of adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (followed by self-sampling for the non-adherent) - SOC+SS (Other): CCS screening according to the standard of care (sample collected by a health professional). Participants not adhering will be subsequently invited to perform self-sampling for screening.
  When considering only the initial use of the SOC for CCS, this corresponds to arm type "active comparator". When considering the use of the SOC, followed by SS for participants not adhering to CCS according to the SOC, this corresponds to arm type "experimental".
  Interventions: Other: Invitation of all participants to CCS according to the standard of care (active comparator); Other: Invitation of all participants to CCS according to the standard of care, followed by invitation of those non-adherent to CCS through self-sampling
- Self-sampling (followed by the standard of care for the non-adherent) - SS+SOC (Experimental): CCS screening by self-sampling. Participants not adhering will be subsequently invited for screening according to the standard of care (sample collected by a health professional).
  Interventions: Other: Invitation of all participants to CCS through self-sampling; Other: Invitation of all participants to CCS through self-sampling, followed by invitation of those non-adherent to CCS according to the standard of care
- Choice (2x) between CCS through sample collected by health professional and self sampling - CHOICEx2 (Experimental): Participants will be asked for their preference for CCS through sample collected by a health professional or by self-sampling, and will undergo CCS accordingly. Those not adhering will be invited again to choose between one of the two methods of CCS.
  Interventions: Other: Invitation of all participants to CCS, asking them to choose between self-sampling and the standard of care; Other: Invitation of all participants to CCS, asking them to choose between self-sampling and the standard of care; this mode of invitation is repeated when participants do not adhere to the first invitation

INTERVENTIONS:
Other: Invitation of all participants to CCS according to the standard of care (active comparator) — Invitation of all participants to CCS according to the standard of care
  Other Names: SOC
  Arms: Standard of care (followed by self-sampling for the non-adherent) - SOC+SS
Other: Invitation of all participants to CCS through self-sampling — A self-sampling kit mailed to the participants, with a prepaid envelope for returning them after sample collection. Participants may also return the kits by depositing them in a container that will be available in their Health Care Center.
  The invitation for CCS through self-sampling is accompanied by written instructions, SMS reminders and navigation support (dedicated telephone line, WhatsApp, website)
  Other Names: SS; Evalyn Brush
  Arms: Self-sampling (followed by the standard of care for the non-adherent) - SS+SOC
Other: Invitation of all participants to CCS, asking them to choose between self-sampling and the standard of care — In a telephone contact, prompted by an SMS, participants will be given the opportunity to schedule CCS according to the standard of care or to ask for a self-sampling kit to be mailed to them. Depending on their choice, the procedure will be similar to what is described for arm SOC or for arm SS, as applicable
  Other Names: CHOICE
  Arms: Choice (2x) between CCS through sample collected by health professional and self sampling - CHOICEx2
Other: Invitation of all participants to CCS according to the standard of care, followed by invitation of those non-adherent to CCS through self-sampling — Participants not adhering to CCS after the first invitation (SOC) will be additionally invited for CCS screening through self-sampling (as in SS)
  Other Names: SOC+SS
  Arms: Standard of care (followed by self-sampling for the non-adherent) - SOC+SS
Other: Invitation of all participants to CCS through self-sampling, followed by invitation of those non-adherent to CCS according to the standard of care — Participants not adhering to CCS after the first invitation for self-sampling (SS) will be additionally invited for CCS screening according to the standard of care (as in SOC)
  Other Names: SS+SOC
  Arms: Self-sampling (followed by the standard of care for the non-adherent) - SS+SOC
Other: Invitation of all participants to CCS, asking them to choose between self-sampling and the standard of care; this mode of invitation is repeated when participants do not adhere to the first invitation — Participants not adhering to CCS after a first invitation for screening through a method of their choice (CHOICE) will be invited again, also being given the opportunity to choose between the standard of care or self-sampling (as in the first CHOICE invitation). Depending on the participants' choice, the procedure will be similar to what is described for arm SOC or for arm SS, as applicable, both in the first and in the second CHOICE invitations
  Other Names: CHOICEx2
  Arms: Choice (2x) between CCS through sample collected by health professional and self sampling - CHOICEx2

SUMMARY:
Cervical cancer screening (CCS) is important to prevent and control cervical cancer (CC). In Portugal, CCS starts with the assessment of the presence of Human Papillomavirus (HPV) in cervical-vaginal samples, collected by a health professional. However, self-sampling (self-collection of vaginal samples by the participants in CCS), is being considered in several settings, aiming to improve participation in CCS, while also exploring its potential to reduce costs.

The goal of this study is to learn how self-sampling could be introduced in the CCS program in Portugal, by testing different strategies to combine the self-collection of samples with the collection of samples by a health professional, which is currently the standard of care.

Researchers will conduct a study comparing the following ways of conducting CCS:

* Sample collection by health professionals - SOC;
* Self-sampling - SS;
* Asking the participants if they prefer to collect their own samples, or to have the samples collected by a health professional, and then proceed as they prefer - CHOICE.

After assessing the adherence to CCS in each of the groups define above, the participants will be given the possibility to participate through a method different from the initially proposed or chosen, as follows:

* SOC will be complemented with invitation for SS;
* SS will be complemented with invitation for the SOC;
* CHOICE participants will be invited again to CHOICE, being given a new opportunity to choose how they prefer to be screened.

This study design allows for comparisons between these groups, to understand how using these strategies alone and complementarily works, and also for comparisons within each group, to understand how one strategy being used on the top of the previous may contribute to increase adherence to screening. The researchers will additionally collect information of the adherence to CCS in the year before the study is conducted, to be used as an additional benchmark.

For a better understanding on the potential barriers and facilitators to incorporating self-sampling in the CCS program, this study will also comprise interviews with the health professionals involved in the study, as well as with females eligible for screening who had been invited to participate.

Depending on the results of HPV testing and complementary cytological evaluations, participants may be referred for further assessment, according to the standard of care in the Portuguese National Health Service. This study will address the possibility of improving the yielding of the referral for further assessment, by testing, in parallel to the current standard of care, a method that is expected to contribute to reducing the number of referrals of false-positives.

Therefore, this study is expected to provide evidence based on different methods of assessment, showing the extent to which SS may contribute to improve adherence do CCS, and testing new methods that may reduce the referral of false-positives for further assessment.

DETAILED DESCRIPTION:
Vaccination against human papillomavirus (HPV) is highly effective and is expected to reduce substantially the burden of cervical cancer (CC), but cervical cancer screening (CCS) remains necessary for females who were not covered by the vaccination plans, those who remain non-adherent to vaccination, and for early detection of the cervical lesions not prevented by the vaccine. However, the sustainability of CCS programs will be challenged by the expectedly dramatic reduction in frequency of cervical precancerous lesions. A paradigm shift for CCS programs, towards a substantial improvement of efficiency, and ability to reach those more in need of screening, is essential to maintain their cost-effectiveness. We will implement a state-of-the-art approach to population-based CCS, with potential to broaden screening coverage, lower costs and increase efficiency, compared to the current standard of care, by including self-sampling and state-of-the-art molecular methods for triage.

The investigation is based on a pragmatic parallel cluster randomized controlled trial (RCT), including nearly 6,000 participants (2,000 in each arm), implemented at Local Health Unit Gaia e Espinho (ULSGE) in collaboration with the Research Center of Portuguese Institute of Oncology of Porto (CI-IPOP). Family doctors will be randomly allocated to one of the three study arms, and all females from their lists of patients who are eligible for screening, as defined by the current guidelines for the organized screening program, will be invited.

CCS screening will be based on high-risk HPV (HrHPV) testing, according to the Portuguese CCS program. Referral to colposcopy will follow the standard of care (based on HrHPV and liquid based cytology [LBC]), regardless of the strategy used for CCS; females testing non-HPV16/18 HrHPV-positive in self-sampling will undergo a new sample collection by a health professional, so that a LBC evaluation can be performed to support the decision of referral to colposcopy, as defined by the standard of care. Deoxyribonucleic acid (DNA) methylation will be conducted in parallel.

Intention to treat analysis will be the primary strategy of analysis for comparison between the groups, based on crude comparisons, or controlling for confounding through multivariable binary logistic regression, when an imbalance between the distribution of confounders between study arms is observed. Methylation accuracy estimates will be computed with 95% confidence intervals. The cutoffs for each biomarker will be those defined in our previous studies.

The sample size was defined to address the primary objectives that involve the comparison of study arms, with a 1:1:1 allocation ratio, considering a statistical power of 90% and a design effect of 1.1 (assuming an average cluster size of 50 and an intracluster correlation coefficient of 0.002). For a non-inferiority hypothesis, considering an alpha (one-sided) of 5% and assuming an adherence of 50% and a non-inferiority margin of 5%, a sample of 5,700 females is needed.

Family doctors from a total of 10 to 20 primary health care units are expected to be enrolled to achieve the sample size needed, depending on the adherence of the medical doctors and the number of eligible females in their lists of patients.

The study will be initially implemented in 2 to 3 primary health care units, to achieve an expected sample of at least 600 participants, for piloting and adjustment of the overall sample size based on the empirical data on the proportions of adherent females in each arm.

The assessment of the adherence according to the different strategies to incorporate self-sampling in the CCS program will be complemented by a qualitative study to assess barriers and facilitators to the implementation of CCS and adherence to CCS in different formats. This will involve the family doctors who have collaborated in the study and females selected among those invited for screening in the different study arms, based on focus groups and individual semi-structured interviews.

Also, a quantitative assessment of the invited females experiences with CCS within the study and determinants of adherence will be conducted on a subsample including approximately 10% of the invited females, who will be asked to answer a structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Females fulfilling the eligibility criteria for CCS, as defined by the current guidelines for the organized screening program in Portugal.

Exclusion Criteria:

* Not having a Portuguese mobile phone number or a Portuguese address available in the clinical/administrative records of the primary healthcare units;
* Any of the exclusion criteria for CCS, as defined by the current guidelines for the organized screening program in Portugal.

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5700 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to screening, after the first invitation for CCS in the study | 45 days after first scheduling/invitation
  Proportion of invited females, in each arm, who adhere after the first scheduling/invitation (SOC, SS or CHOICE)
Adherence to CCS, after two invitations for screening in the study | 45 days after first scheduling/invitation or 45 days after the second scheduling/invitation (for those not adhering to the first scheduling/invitation within 45 days)
  Proportion of invited females, in each arm, who adhere after the second scheduling/invitation (SOC+SS, SS+SOC or CHOICEx2)
Performance of DNA methylation markers for high-grade squamous intraepithelial lesions or worse (HSIL+) detection | 45 days after cytological or histological results, as applicable
  Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of methylation analysis for detection of high-grade squamous intraepithelial lesions or worse (HSIL+), using the cytological triage results and the histological results as gold-standard

SECONDARY OUTCOMES:
Identification of barriers and facilitators to the implementation and participation in CCS | 90 days after the last invitation for CCS in the study
  Perception of medical doctors and females eligible for CCS regarding barriers and facilitators to the implementation and participation in CCS, assessed through qualitative research, based on focus groups and semi-structured interviews
Proportion of HPV infection, overall and for each genotype tested | 45 days after first scheduling/invitation or 45 days after the second scheduling/invitation (for those not adhering to the first scheduling/invitation within 45 days)
  Proportion of invited and of adherent females, in each arm, testing positive for HPV infection and for the different genotypes tested, after the first invitation/scheduling (SOC, SS or CHOICE) and after the second scheduling/invitation (SOC+SS, SS+SOC or CHOICEx2)
Adherence to follow-up appointments (%), overall and among participants referred for follow-up | 45 days after the appointment date
  Proportion of invited and of HPV-positive (eligible for referral according to the guidelines) females, in each arm, referred for follow-up appointments, after the first invitation/scheduling (SOC, SS or CHOICE) and after the second scheduling/invitation (SOC+SS, SS+SOC or CHOICEx2)
Variation in adherence and HPV test result outcomes between the first and the second invitation for screening | 45 days after first scheduling/invitation or 45 days after the second scheduling/invitation (for those not adhering to the first scheduling/invitation within 45 days)
  Variation in all adherence and HPV test result outcomes between the first and the second invitation for screening (before-after comparison), in each arm
Variation in adherence from the previous year to the study period | 45 days after first scheduling/invitation or 45 days after the second scheduling/invitation (for those not adhering to the first scheduling/invitation within 45 days)
  Before-after comparison of the proportion of adherence during the study with the proportion of adherence among the patients from each participating medical doctor in the previous year (aggregated data), overall in each arm, and by medical doctor
Subgroup analyses of all comparisons of adherence between groups | 45 days after first scheduling/invitation or 45 days after the second scheduling/invitation (for those not adhering to the first scheduling/invitation within 45 days)
  Stratified analyses of the adherence outcomes, according to age groups, deprivation index of the place of residence, primary health care unit, organization model of the primary healthcare units (USFA, USFB or UCSP) and CCS history
Subgroup analyses of DNA methylation accuracy outcomes, according to the adherence to self-sampling and to the standard of care | 45 days after cytological or histological results, as applicable
  Stratified analyses of the accuracy outcomes, overall and in each arm
Characterization of the experience with CCS and determinants of adherence | 120 days after the last invitation for CCS in the study
  The experience of females invited to CCS as well as the determinants of adherence will be assessed through an observational design based on a subsample of females invites to the study, quantified using descriptive statistics and crude and adjusted odds ratios

OTHER OUTCOMES:
Process indicators | Up to 45 days after first scheduling/invitation or up to 45 days after the second scheduling/invitation (for those not adhering to the first scheduling/invitation within 45 days)
  Variation of adherence over time since invitation/scheduling; contacts with the help-line and their timing and contents; returned letters/messages due to incorrect address/contact number; missed CCS appointments; rescheduled CCS appointments; samples inadequate for analysis; time spent in the different tasks

CONTACTS AND LOCATIONS:
Overall Officials: Nuno Lunet, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Unidade Local de Saúde Gaia e Espinho, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: No